CLINICAL TRIAL: NCT07034976
Title: Randomized, Controlled Trial to Evaluate the Efficacy of Non-ablative Radiofrequency Combined With Pelvic Floor Muscle Training on Symptoms of Genitourinary Syndrome of Menopause in Breast Cancer Survivors
Brief Title: Efficacy of Non-ablative Radiofrequency Combined With Pelvic Floor Muscle Training for Genitourinary Syndrome of Menopause in Breast Cancer Survivors (RF-SGM)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Collaborators: Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Principal Investigator, Irene Lázaro Navas, PhD Physiotherapist, Department of Rehabilitation Medicine, Hospital Universitario Ramón y Cajal, Hospital Universitario Ramon y Cajal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 069/25; IMP24_B01 (Other Grant/Funding Number: Biomedical Research Foundation of Ramón y Cajal University Hospital (FIBio-HRC))
Record Dates: First submitted 2025-05-27; First posted 2025-06-24 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-07

CONDITIONS: Genitourinary Syndrome of Menopause (GSM); Breast Cancer
Keywords: genitourinary syndrome of menopause; vaginal atrophy; vaginal dryness; breast cancer survivors; non-ablative radiofrequency; pelvic floor muscle training; physiotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessors will be blinded to group allocation. In addition, the independent statistician responsible for data analysis will remain blinded until the database is locked. Only the treating physiotherapists and the study coordinator will have access to the randomization list
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Non-ablative Radiofrequency + Pelvic-Floor Muscle Training (Experimental): Participants in this group will receive non-ablative monopolar capacitive radiofrequency therapy combined with pelvic-floor muscle training guided by biofeedback.
  Interventions: Device: Active Radiofrequency (Capenergy C500 UpGradeC200)
- Sham Radiofrequency + Pelvic-Floor Muscle Training (Sham Comparator): Participants in this group will receive sham radiofrequency treatment combined with pelvic-floor muscle training guided by biofeedback.
  Interventions: Device: Sham Radiofrequency (Capenergy C500 UpGrade C200 - Placebo Mode)

INTERVENTIONS:
Device: Active Radiofrequency (Capenergy C500 UpGradeC200) — Non-ablative radiofrequency is applied using a Capenergy C500 device at a target tissue temperature of ≤ 45 °C, once a week for 6 consecutive weeks. Treatment is delivered through two channels simultaneously: a capacitive plate placed on the suprapubic area and an intracavitary vaginal probe. Each session lasts 20 minutes and is followed by 20 minutes of pelvic-floor muscle training guided by biofeedback. Participants will also follow a progressive home exercise programme and record adherence and events.
  In addition, all participants will receive education on pelvic-floor anatomy and function, underlying mechanisms of pain after breast cancer, bladder and bowel retraining, respiratory pattern re-education, and-if interested-information on sexual health.
  Arms: Active Non-ablative Radiofrequency + Pelvic-Floor Muscle Training
Device: Sham Radiofrequency (Capenergy C500 UpGrade C200 - Placebo Mode) — Participants will receive one session per week for 6 weeks of sham (placebo) radiofrequency using the Capenergy C500 in Placebo Mode (no temperature increase), designed to simulate active treatment. The screen will display a simulated "delivered energy" value; temperature and energy readings will be hidden; LED indicators will activate sequentially; and a suprapubic capacitive plate and intracavitary probe will be used with the same protocol as in the intervention group. This will be followed by 20 minutes of pelvic-floor muscle training guided by biofeedback, identical to the intervention group. Participants will also follow a progressive home exercise programme and record adherence and events. All participants will receive education on pelvic-floor function, pain mechanisms after breast cancer, bladder/bowel retraining, breathing pattern correction, and-if interested-sexual health.
  Arms: Sham Radiofrequency + Pelvic-Floor Muscle Training

SUMMARY:
The goal of this clinical trial is to find out whether non-ablative radiofrequency (RF) applied together with pelvic-floor muscle exercises can ease vaginal dryness and other symptoms of genitourinary syndrome of menopause (GSM) in women aged 18-75 years who have survived breast cancer and currently experience those symptoms.

The main questions it aims to answer are:

Does the combination of RF + exercise lower the 0-to-10 vaginal-dryness score more than sham (inactive) RF + exercise at 6 weeks (end of treatment) and 3 months?

What other changes (pain during intercourse, Vaginal Health Index, urinary and sexual function, pelvic-floor strength, overall satisfaction) are seen in each group?

Researchers will compare six sessions of active RF with six sessions of sham (inactive) RF to see whether the active treatment works better.

Participants will:

Visit the hospital once a week for 6 weeks. Each visit includes about 20 minutes of intra-/extra-vaginal RF (or sham) and 20 minutes of guided pelvic-floor training whose content is adapted and progressed throughout the study.

Carry out a structured, progressive home-exercise programme, recording any discomfort in a diary.

Complete questionnaires and tests at baseline, after session 6, and 3 months later.

ELIGIBILITY:
Inclusion Criteria:

* Women who are breast cancer survivors and clinically confirmed to be disease-free by their physician.
* Amenorrhea for more than 12 months and vaginal pH ≥ 5, with symptoms related to genitourinary syndrome of menopause (GSM), as diagnosed by a physician. Symptoms must be bothersome and not better explained by another clinical condition.
* Negative urine culture at baseline.
* Moderate to severe vaginal dryness, defined as a score > 4 on the Numeric Rating Scale (NRS 0-10)

Exclusion Criteria:

* Age over 75 years.
* Current or past diagnosis of any cancer other than breast cancer.
* Pelvic surgery, chemotherapy, or radiotherapy in the past 3 months.
* Use of local estrogen therapy within the past month.
* Active genital infections.
* Diagnosis of HIV infection or severe immunosuppression.
* Presence of pacemakers, metallic implants, or electromagnetic devices.
* Coagulation disorders or current use of anticoagulants.
* Pelvic organ prolapse stage > III (POP-Q classification).
* Unexplained abnormal vaginal bleeding.
* History of pelvic anti-incontinence surgery, with or without mesh.
* Inflammatory dermatoses of the vulva.
* Pelvic-floor muscle strength score of 0/5 on the Modified Oxford Scale.
* Nickel allergy.
* Previous treatment with radiofrequency in the pelvic or genital area.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Subjective sensation of vaginal dryness | T0 (baseline, before intervention); T1 (immediately after completing the intervention); T2 (3 months after T1)
  Measured using a 0-10 Numeric Rating Scale (NRS), where 0 indicates "no dryness" and 10 indicates "maximum dryness". The NRS is a self-reported, single-item scale commonly used for subjective symptom intensity.

SECONDARY OUTCOMES:
Subjective sensation of pain during sexual activity (NRS 0-10) | T0 (baseline, before intervention); T1 (immediately after completing the intervention); T2 (3 months after T1)
  Measured using a 0-10 Numeric Rating Scale (NRS), where 0 indicates "no pain" and 10 indicates "maximum pain during sexual activity". The NRS is a self-reported, single-item scale commonly used for subjective symptom intensity.
Subjective sensation of vaginal itching (NRS 0-10) | T0 (baseline, before intervention); T1 (immediately after completing the intervention); T2 (3 months after T1)
  Measured using a 0-10 Numeric Rating Scale (NRS), where 0 indicates "no itching" and 10 indicates "maximum itching". The NRS is a self-reported, single-item scale commonly used for subjective symptom intensity.
Vaginal Health Index Score | T0 (baseline, before intervention); T1 (immediately after completing the intervention); T2 (3 months after T1)
  The Vaginal Health Index Score assesses five parameters (elasticity, secretions, epithelial integrity, moisture, and pH), each rated from 1 to 5. The total score ranges from 5 (worst condition) to 25 (optimal vaginal health).
Female Sexual Function Index total score | T0 (baseline, before intervention); T1 (immediately after completing the intervention); T2 (3 months after T1)
  The FSFI is a 19-item self-reported questionnaire evaluating six domains: desire, arousal, lubrication, orgasm, satisfaction, and pain. Total scores range from 2 to 36. A score below 26.55 is considered indicative of sexual dysfunction based on established clinical cutoffs.
Vaginal pH level | T0 (baseline, before intervention); T1 (immediately after completing the intervention); T2 (3 months after T1)
  The pH will be quantified using MColorpHast™ pH indicator strips (0-14 range, Merck®). The strip will be placed directly on the right lateral vaginal wall for a few seconds, and the result will be determined by comparing the colour to the manufacturer's reference scale. Higher pH values are typically associated with hypoestrogenic states and genitourinary symptoms of menopause
Pelvic organ support parameters measured by POP-Q system | T0 (baseline, before intervention); T2 (3 months after T1)
  Pelvic anatomy will be assessed using the Pelvic Organ Prolapse Quantification (POP-Q) system, with the patient in gynecological position and using a speculum. The following parameters will be recorded: genital hiatus (GH), perineal body (PB), total vaginal length (TVL), and reference points Aa, Ba, C, D, Ap, and Bp.
International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF total score) | T0 (baseline, before intervention); T1 (immediately after completing the intervention); T2 (3 months after T1)
  The ICIQ-SF is a self-reported questionnaire assessing the frequency, severity, and impact of urinary incontinence. Scores range from 0 to 21, with higher scores indicating greater severity.
ICIQ-FLUTS | T0 (baseline, before intervention); T1 (immediately after completing the intervention); T2 (3 months after T1)
  The ICIQ-FLUTS (International Consultation on Incontinence Questionnaire - Female Lower Urinary Tract Symptoms) is a self-administered questionnaire designed to evaluate female lower urinary tract symptoms (LUTS) and their impact on quality of life. It consists of 12 items grouped into three independent domains: storage symptoms, voiding symptoms, and incontinence symptoms. Each item assesses the presence and perceived severity of the symptom
Pelvic-floor muscle strength (Modified Oxford Scale, 0-5) | T0 (baseline, before intervention); T1 (immediately after completing the intervention); T2 (3 months after T1)
  Assessed by vaginal palpation using the Modified Oxford Scale, which rates voluntary pelvic-floor muscle contraction from 0 (no contraction) to 5 (strong contraction). This is a validated, clinician-administered tool.
Pelvic-floor muscle activity measured by surface electromyography (μV) | T0 (baseline, before intervention); T1 (immediately after completing the intervention); T2 (3 months after T1)
  Pelvic-floor muscle activation is measured using surface electromyography (sEMG) with an intracavitary Periform® vaginal probe. The outcome is expressed in microvolts (μV) and reflects the neuromuscular response of the pelvic floor during both contraction and resting phases. For each participant, the final value will be calculated as the mean of three voluntary contractions, with 10-second rest intervals between contractions
Subjective global impression of improvement (7-point Likert scale) | T1 (immediately after completing the intervention); T2 (3 months after T1)
  Participants will be asked to rate their overall perception of improvement in symptoms after the intervention using a 7-point Likert scale, specifically designed for this study and based on the Patient Global Impression of Change (PGIC). The scale ranges from 1 ("very much improved") to 7 ("very much worse"), reflecting the participant's subjective global impression of improvement compared to their baseline condition.
Incidence of adverse events related to the intervention | T1 (immediately after completing the intervention); T2 (3 months after T1)
  Any unexpected or undesired sign, symptom, or condition temporally associated with the intervention will be recorded
Adherence to prescribed home pelvic-floor training | T1 (immediately after completing the intervention); T2 (3 months after T1)
  Measured through a self-reported diary where participants record the frequency and completion of home-based pelvic-floor exercises. Adherence is expressed as a percentage of the total prescribed sessions completed.
Local recurrence of breast cancer at 12 months | 12 months after T1
  Oncological follow-up will document any confirmed local breast cancer recurrence occurring within 12 months of completing the intervention.
Participant's belief regarding group allocation (intervention vs. placebo) | T1 (immediately after completing the intervention)
  At the end of the intervention, participants will be asked whether they believe they received the active treatment or the placebo treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Ramón y Cajal, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided
The decision to share individual participant data (IPD) has not been finalized. Any future data sharing will follow applicable ethical, legal, and institutional guidelines.